CLINICAL TRIAL: NCT03180073
Title: Prevalence and Significance of Bradycardic Arrhythmias and Conduction Abnormalities Among Patients With Severe Aortic Stenosis Before and After Transcatheter Aortic Valve Replacement Using Extended Heart Rhythm Recording (Brady-TAVR Study)
Brief Title: Conduction Abnormalities With Severe Aortic Stenosis Before and After Transcatheter Aortic Valve Replacement
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Khaldoun Tarakji, Principal Investigator, The Cleveland Clinic
Other Study IDs: 17-086
Record Dates: First submitted 2017-05-09; First posted 2017-06-08 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ziopatch Pre discharge — Ziopatch applied 2 weeks prior to procedure
Diagnostic Test: Ziopatch at Discharge — Ziopatch applied at discharge from hospital to be worn for 2 weeks
Diagnostic Test: Ziopatch at 2 months — Ziopatch applied 2 months from procedure to be worn for 2 weeks

SUMMARY:
Most of the conduction abnormalities with TAVR are usually detected during the procedure or during the following days of observation. Little is known about the prevalence and timing of any conduction abnormalities that exist before (other than standard ECG) or after through long term cardiac monitoring.

DETAILED DESCRIPTION:
Each subject who fulfills the inclusion/exclusion criteria will be provided with Zio patch for 2 weeks before TAVR. Immediately after the procedure, patients will be admitted per TAVR protocol and will be on telemetry. Data about their ECGs and any arrhythmias will be collected.

Upon discharge, patients will be provided with another Zio patch for 2 weeks. At the 2-3 months follow up, subjects will be provided with a third Zio patch for 2 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 and <90 years old
2. Able to provide informed consent
3. Willing to follow up at Cleveland Clinic (per TAVR protocol)

Exclusion Criteria:

1. Prior CIED (Pacemaker or defibrillator)
2. Unable to provide consent
3. Unable to follow up at Cleveland Clinic per TAVR protocol

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients to be scheduled for TAVR without preexisting Cardiac Implantable Electronic Device (CIED) can be screen and enrolled
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2020-12-23 (Actual); Study Completion 2020-12-23 (Actual)

PRIMARY OUTCOMES:
Need for Pacemaker post TAVR | 2 months prior to TAVR
  the prevalence of brady arrhythmia (Sinus brady, Sinus Pauses, AV Block, Bundle Branch Block) among patients with severe aortic stenosis who undergo TAVR using an extended cardiac rhythm monitor (Zio Patch) and determine if the brady arrhythmias predict the need for a pacemaker.

SECONDARY OUTCOMES:
Prevalence of in hospital brady arrhythmia post TAVR | 72 hours post TAVR
  the prevalence of brady arrhythmia (Sinus brady, Sinus pause, AV block, Bundle branch block) using hospital telemetry data
Prevalence of brady arrhythmia after discharge from hospital post TAVR | 3 weeks post discharge
  the prevalence of brady arrhythmia (Sinus brady, Sinus pauses, AV block, Bundle branch block) using extended cardiac rhythm monitor (Zio Patch)
Prevalence of delayed brady arrhythmia post TAVR | 2 months post TAVR
  the prevalence of brady arrhythmia using extended cardiac rhythm Assess the prevalence of brady arrhythmia (Sinus brady, Sinus Pause, AV block, Bundle branch block) using extended cardiac rhythm monitor (Zio Patch)

CONTACTS AND LOCATIONS:
Overall Officials: Khaldoun Tarakji, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tarakji KG, Patel D, Krishnaswamy A, Hussein A, Saliba W, Wilkoff BL, Wolski K, Svensson L, Wazni OM, Kapadia SR. Bradyarrhythmias detected by extended rhythm recording in patients undergoing transcatheter aortic valve replacement (Brady-TAVR Study). Heart Rhythm. 2022 Mar;19(3):381-388. doi: 10.1016/j.hrthm.2021.11.020. Epub 2021 Nov 18. PMID 34801735